CLINICAL TRIAL: NCT04159688
Title: Imaging Glutamate Release From Alcohol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000026672; 1K01AA024788-01A1 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol Challenge (Experimental): Alcohol Challenge, oral, targeting BAL of 60 mg/dL, Given once
  Interventions: Drug: Alcohol

INTERVENTIONS:
Drug: Alcohol — Alcohol Challenge

SUMMARY:
The goal of this research project is to determine the sensitivity of PET radioligands specific for targets in the glutamate system to an alcohol challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 21-55 years
2. Willing and able to give voluntary written informed consent
3. Able to read and write English and communicate effectively with the investigators, and comply with all study requirements, restrictions, and directions of the clinic staff
4. Moderate Drinkers will report consuming alcohol on at least one occasion in the past three months that would result in an estimated blood alcohol level greater than 100 mg/dl but not meet DSM-5 criteria for AUD. This is to ensure that subjects have prior drinking exposure consistent with levels proposed in this study. Prospective subjects will be asked to recall the heaviest two days of drinking in the previous three months. Using this information, approximate BAC will be calculated for those prior episodes.
5. Medically healthy upon physical examination and laboratory testing.

Exclusion Criteria:

1. Individuals whom the investigators deem may not be able to comply with alcohol abstinence for 48 hours prior to study day.
2. Current significant medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology.
3. History of or current neurological or significant psychiatric disorder such as schizophrenia or bipolar disorder (DSM-5 Axis 1).
4. Other substance use disorder with the exception of nicotine dependence in smokers as assessed with the SCID or positive urine screen for drugs of abuse.
5. Participants with any significant current medical conditions that would contraindicate the consumption of alcohol, such as history of neurological trauma or diseases, seizures, delirium or hallucinations, hepatic, or other unstable medical conditions.
6. Current suicidal or homicidal intent or behavior, or history of suicidal or homicidal behavior.
7. No barbiturates or other known microsomal enzyme induces or inhibitors in the past month.
8. History of significant head trauma.
9. Women who are pregnant or nursing or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD).
10. Regular or current significant use of any prescription, herbal or illegal psychotropic medications (e.g., antidepressants, antipsychotics, anxiolytics, ecstasy) in the past 6 mo, with no current illegal drug use confirmed by urine toxicology (except for cocaine and marijuana when relevant).
11. Have MRI-incompatible implants and other contraindications for MRI, such as a pacemaker, artificial joints, non-removable body piercings, claustrophobia, etc.
12. Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
13. Subjects with current, past or anticipated exposure to radiation in the work place within one year of proposed research PET scans.
14. Subjects with history of IV drug use which would prevent venous access for PET tracer injection.
15. Blood donation within eight weeks of the start of the study
16. History of blooding disorder or currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ansel T Hillmer, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol Challenge
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alcohol Challenge
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Alcohol-induced Change in Receptor Availability
Description: The percent change in receptor availability will be measured from the PET data. Since this project is for basic science it is not known whether positive values are better or worse outcome.
Time Frame: Baseline and within 2 hours of challenge
Measure: Mean (Full Range); unit: percentage change of BP_ND
Arm/Group | Alcohol Challenge
Number analyzed (Participants) | 7
percentage change of BP_ND | -9.1 [-11.2 to -6.6]

ADVERSE EVENTS:
Time Frame: 2 Months
Arm/Group | Alcohol Challenge
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT04159688/Prot_SAP_000.pdf